CLINICAL TRIAL: NCT06971809
Title: Efficacy of a Multi-modal Pain Resilience Approach to Chronic Low Back Pain
Brief Title: Pain Resilience for Low Back Pain.
Acronym: Resilience
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Pain Science Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #180-23
Record Dates: First submitted 2025-03-06; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Low Back Pain (CLBP)

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fear group (Active Comparator): This intervention addresses the negative valence system to decrease fear and threat.
  Interventions: Behavioral: Pain education
- Strengths group (Active Comparator): This group addresses the positive valance system for reward learning
  Interventions: Behavioral: Pain resilience

INTERVENTIONS:
Behavioral: Pain resilience — A strengths-based approach to pain recovery
  Arms: Strengths group
Behavioral: Pain education — A health literacy approach
  Arms: Fear group

SUMMARY:
Chronic pain affects about 20% of adults in the U.S. and can lead to serious personal, social, and economic challenges. It is often treated with medications, including opioids, which carry risks of dependence. While pain education (PE) helps people better understand their pain and may reduce symptoms, it generally has only modest effects when used alone.

The purpose of this study is to explore whether combining pain education with other treatments-such as physical therapy, cognitive behavioral techniques, and healthy lifestyle strategies-in a multi-modal resilience approach can offer greater benefits. The study aims to answer the following question:

Can a combined, whole-person approach improve outcomes in people with chronic pain more effectively than pain education alone?

DETAILED DESCRIPTION:
Chronic pain is pain that lasts beyond the typical healing duration, and is typically defined as lasting for at least 3-6 months. Approximately 20% of the adult U.S. population experiences chronic pain. There are a variety of risk factors for developing chronic pain. Female sex, older age, living in poverty, having chronic health conditions or a disability and being a veteran are among the risk factors for chronic pain. Chronic pain impacts quality of life as well as worker productivity. Chronic pain presents an economic burden beyond absenteeism and lost wages and costs the healthcare system upwards of $300 billion for a range of services including medication for pain management, surgeries, and disability compensation. Additionally, opioid prescription for chronic pain is a primary driver of opioid use disorder. Teaching those with chronic pain how to effectively manage their pain can improve quality of life and reduce the risk of developing dependency on opioid medication.

The non-pharmacologic and non-invasive treatment of chronic pain includes physical therapy, cognitive behavioral techniques, and strategies for promoting a healthy lifestyle. Pain education (PE) has been advocated as a methodology to reduce chronic pain. PE teaches that pain is not simply the result of tissue damage. Rather, the foundation of PE is education about the factors that can contribute to pain such as emotions, beliefs, and past experiences.4 However, PE is a singular modality that produces small effects. A multi-modal resilience approach model may produce larger effects.

ELIGIBILITY:
Inclusion Criteria

* Adults experiencing chronic pain of any diagnosis for a duration of at least 6 months.
* Ability to read and understand English.

Exclusion Criteria

* Experiencing acute pain related to a recent injury or pain lasting less than 6 months.
* Inability to read or understand English.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | 90 days
  Pain intensity will be measured by the Defense of Veterans Pain Rating Scale. This is a numerical scale with descriptors
  0 = No pain
  1. = Hardly noticeable pain
  2. = Noticeable pain, but does not interfere with activities
  3. = Somewhat distracting pain
  4. = Distracting pain, but does not affect normal activities
  5. = Pain interrupts some activities
  6. = Hard to ignore pain, avoidance of daily activities
  7. = Pain is the main focus of attention, prevents daily activities
  8. = Awful pain, difficult to do anything
  9. = Unbearable pain, cannot do anything
  10. = As bad as pain can be, nothing else matters

SECONDARY OUTCOMES:
Optimal Screening for Prediction of Referral and Outcome-Yellow Flag (OSPRO-YF) | 90 days
  The Optimal Screening for Prediction of Referral and Outcome-Yellow Flag (OSPRO-YF) is an assessment tool designed to help orthopedic physical therapy clinicians screen patients and clients for psychosocial distress. Test items assess depression, anxiety, kinesiophobia, anger, fear-avoidance beliefs, catastrophizing, self-efficacy, and pain acceptance. As OSPRO-YF summarizes 11 psychological questionnaires, it is not scored like a conventional screening tool. Quartile scores are used instead of cutoff scores for consistency and assessment. Scores that are in the top quartile (top 25%) for negative psychological questionnaires (Negative Mood and Fear Avoidance questionnaires) Scores that are in the bottom quartile (bottom 25%) for positive psychological questionnaires (Positive Affect/Coping questionnaires).

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Palombero, PhD, Study Director — Widener University
Locations (1):
- Integrative Pain Science Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol will be shared.
Supporting Information: Study Protocol
Time Frame: June 2025-June 2026
Access Criteria: The study protocol will be shared with qualified investigators whose aims address sound scientific questions related to pain management. Interested parties must submit a proposal outlining their planned analyses, which will be reviewed before approval. Upon acceptance, a use agreement must be signed, and data will be shared via a secure platform.
URL: http://www.integrativepainscienceinstitute.com